CLINICAL TRIAL: NCT04682691
Title: Comparison of the Effect of Metoclopramide Versus Erythromycin on Gastric Residual Volume
Brief Title: Effect of Metoclopramide Versus Erythromycin on on Gastric Residual Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS-381-2020
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Gastric Residual Volume
Keywords: Erythromycin; Gastric Emptying; Metoclopramide; Ultrasonography
MeSH Terms: interventions — Erythromycin; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group (C) (Sham Comparator): will be receive flavored water in total volume 15 ml
  Interventions: Dietary Supplement: naturally flavored water
- Group (M) (Active Comparator): will be receive 10 ml of oral metoclopramide (10mg) + 5 ml of flavored water in total volume 15 ml
  Interventions: Drug: metoclopramide (10mg)
- Group (E) (Active Comparator): will be receive 10 ml of oral Erythromycin (400mg) + 5 ml of flavored water in total volume 15 ml
  Interventions: Drug: Erythromycin (400mg)

INTERVENTIONS:
Drug: Erythromycin (400mg) — oral Erythromycin (400mg)
  Arms: Group (E)
Drug: metoclopramide (10mg) — oral metoclopramide (10mg)
  Arms: Group (M)
Dietary Supplement: naturally flavored water — naturally flavored water
  Arms: Group (C)

SUMMARY:
In emergencies, it may be necessary to anaesthetize who are not fully starved and consequently at risk of pulmonary aspiration. Pregnancy are recognized to be at increased risk of aspiration compared with non-pregnancy. Prokinetic agents such as metoclopramide can be used to reduce GRV. Metoclopramide is widely used as a prokinetic agent in adults and is licensed for premedication in pregnancy, but its use may be limited by its potential for producing extrapyramidal side effects. Erythromycin is an effective prokinetic agent in adults but there is no work examining its use for premedication in pregnancy. This study compared the effects of erythromycin and metoclopramide on GRV in full-term pregnant women

ELIGIBILITY:
Inclusion Criteria:

* Non-laboring pregnant women ≥36 weeks gestational age
* Parturient scheduled for elective caesarian delivery.
* Singleton pregnancy
* Age greater than 18 years
* Having followed institutional fasting guidelines (a minimum of 2 h for clear fluids, 6 h for a light meal, and 8 h for a meal that included fried or fatty food)

  2. Exclusion criteria:
* Refusal of the patient
* Deviation from fasting times
* Patients with empty stomach
* Emergency operation
* Body mass index (BMI) greater than 40 kg/m2
* American Society of Anesthesiologists (ASA) physical status class III, IV.
* Gestational diabetes mellitus
* Multiple gestations
* Patients with polyhydramnios liquor.
* Preeclampsia patients
* Chronic kidney disease patients
* Systemic diseases may cause delayed gastric emptying (eg: myopathies and myasthenia gravis).
* Patients with gastrointestinal diseases such as hiatus hernia, intestinal disease and gastro-oesophageal reflux disease and patients with history of upper gastrointestinal surgeries.
* Patients on antidepressants and monoamine oxidase inhibitors
* Use of other medications known to affect gastric motility or secretions.
* Allergy to macrolide or metoclopramide

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only pregnancy women
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Estimated Gastric volume | UP TO 6 HOURE
  (ml/kg) after a six-hour fast using Roukhomovsky's equation after administration of the study drug.

SECONDARY OUTCOMES:
low-risk stomach six hours after drug administration | up to 6 hours
  number of patient and %
Perlas grading system | UP TO 24 HOURE
  Grade 0 antrum: absent fluid content in both supine and RLD positions Grade 1 antrum: fluid is observed only in the RLD position, but not in the supine position Grade 2 antrum: fluid is observed in both supine and RLD
Evaluation of the risk of aspiration | UP TO 24 HOURE
  residual gastric volume < 1.5 mL/kg
quantitative gastric contents | up to 24 hours
  every one hours estimated GV till ( < 1.5 ml/kg) post-drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Amr wahdan, MD, Principal Investigator — Cairo university , Cairo, Egypt
Locations (1):
- Faculty of Medicine, Cairo University., Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided